CLINICAL TRIAL: NCT03361293
Title: Neuromodulation Augmented Cognitive Remediation to Improve Executive Dysfunction in Fetal Alcohol Spectrum Disorder (FASD)
Brief Title: Cognitive Training and tDCS for Children With FASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2017-26075
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: 1:1 randomized allocation to active tDCS or placebo (sham tDCS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and families will be blinded. The principal investigator will be blinded. The research staff member coordinating the visit will be blinded. The care provider is not involved in the research and is, therefore, blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cognitive Training and Active tDCS (Active Comparator): 5 sessions of computerized cognitive training on tasks of attention, concentration, set-shifting, and memory - plus active tDCS (also 5 sessions).
  Interventions: Device: Active tDCS; Behavioral: Cognitive training
- Cognitive Training and Sham tDCS (Sham Comparator): 5 sessions of computerized cognitive training on tasks of attention, concentration, set-shifting, and memory - plus sham tDCS (also 5 sessions) which consists of "placebo" stimulation with tDCS (ramp-up, but no actual stimulation).
  Interventions: Behavioral: Cognitive training; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active Transcranial Direct Current Stimulation (tDCS) administered with a Neuroelectrics StarStim Enobio cap system (active mode)
  Arms: Cognitive Training and Active tDCS
Behavioral: Cognitive training — BrainHQ Computerized cognitive training
Device: Sham tDCS — Sham Transcranial Direct Current Stimulation (tDCS) administered with a Neuroelectrics StarStim Enobio cap system (sham mode)
  Arms: Cognitive Training and Sham tDCS

SUMMARY:
This is a randomized placebo-controlled trial of cognitive training with transcranial direct current stimulation (tDCS) for children and adolescents (ages 10 - 16 years) with prenatal alcohol exposure (PAE).

DETAILED DESCRIPTION:
Prenatal alcohol exposure (PAE) has profound detrimental effects on brain development and, as a result, has permanent consequences for cognition, learning, and behavior. Individuals with Fetal Alcohol Spectrum Disorders (FASD) commonly have a range of neurocognitive impairments that directly lead to practical problems with learning, attention, working memory, task planning/execution, and decision making, among other areas of functioning. Despite the profound public health burden posed by FASD, there have been very few treatment studies in this population. This study will examine the effects of a cognitive remediation training augmented with tDCS in children and adolescents with PAE. Functional magnetic resonance imaging will be collected to provide preliminary data of brain circuitry changes created by this intervention. The study involves a baseline visit with cognitive testing, MRI, 5 sessions of tDCS (including the baseline visit), and a 6th visit for cognitive testing and MRI. All sessions will be completed within a 28 to 56 day time window.

ELIGIBILITY:
Inclusion Criteria:

* Documented heavy prenatal alcohol exposure (self-report, social service records, or adoption records) and meeting criteria for an associated FASD diagnosis (FAS, partial FAS, or ARND).
* An available parent or legal guardian capable of giving informed consent

Exclusion Criteria:

* Substance abuse in the participant
* Neurological condition or other developmental disorder
* Serious psychiatric disorder known to affect brain functioning and cognitive performance
* Birthweight < 1500 grams
* MRI contraindication
* tDCS contraindication

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wozniak, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boroda E, Krueger AM, Bansal P, Schumacher MJ, Roy AV, Boys CJ, Lim KO, Wozniak JR. A randomized controlled trial of transcranial direct-current stimulation and cognitive training in children with fetal alcohol spectrum disorder. Brain Stimul. 2020 Jul-Aug;13(4):1059-1068. doi: 10.1016/j.brs.2020.04.015. Epub 2020 Apr 28. PMID 32360392

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Started | 20 | 24
Completed | 19 | 19
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 19 | 38
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 2 | 2 | 4
  White | 9 | 11 | 20
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Delis Rating of Executive Functioning (D-REF) [Mean (Standard Deviation); unit: t-score] — The Delis Rating of Executive Functioning (D-REF) contains 60 items rated by the parent to measure the child's executive functioning compared to age-peers. Results are calculated as T-scores, which have a mean of 50 and a standard deviation of 10. Here, we present the scores at study baseline (visit 1), pre-intervention. Greater values reflect greater executive functioning impairment.
  Time Frame: D-REF will be administered at baseline and at the final visit (28 to 56 days after baseline). NOTE that outcome scores are listed in the appropriate section
  t-score | 69.9 (9.0) | 76.3 (11.7) | 72.4 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: BrainHQ Learning Rate
Description: Participants completed a Divided Attention Task during 5 sessions of tDCS. Unit of measure: milliseconds Meaning: lowest threshold reached across trials / fastest reaction time Direction: lower values represent better performance
Time Frame: Learning rate will be computed over 5 sessions of tDCS spanning 28 to 56 days; Each of the 5 tDCS sessions are 46 minutes long. The divided attention task is administered at the end of each tDCS session.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
milliseconds | 867.6 (244.1) | 861.7 (264.2)

2. Secondary Outcome: Change in D-KEFS Verbal Fluency - Letter
Description: The Delis-Kaplan Executive Function System (D-KEFS) cognitive battery measures executive functioning skills. Task performance is in scaled score points based on items generated and errors (range of 1-19 with a mean of 10 and a standard deviation of 3). Here, we present difference scores between session 1 (baseline) and 5 (completion). Greater values represent more change. Positive values represent improvement; negative values represent decline in performance.
Time Frame: D-KEFS will be administered at baseline and at the final visit (28 to 56 days after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
score on a scale | -0.11 (2.05) | -0.05 (1.68)

3. Secondary Outcome: Change in D-KEFS Verbal Fluency - Category
Description: as for outcome 2
Time Frame: D-KEFS will be administered at baseline and at the final visit (28 to 56 days after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
score on a scale | -3.68 (3.93) | -3.42 (3.37)

4. Secondary Outcome: Change in D-KEFS Trail-making - Numbers
Description: as for outcome 2
Time Frame: D-KEFS will be administered at baseline and at the final visit (28 to 56 days after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
score on a scale | 1.11 (3.2) | 1.37 (3.2)

5. Secondary Outcome: Change in D-KEFS Trail-making - Letters
Description: as for outcome 2
Time Frame: D-KEFS will be administered at baseline and at the final visit (28 to 56 days after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
score on a scale | 1.05 (3.29) | -2.95 (3.73)

6. Secondary Outcome: Change in D-KEFS Trail-making - Combined
Description: as for outcome 2
Time Frame: D-KEFS will be administered at baseline and at the final visit (28 to 56 days after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
score on a scale | -1.16 (6.24) | -2.05 (6.18)

7. Secondary Outcome: Delis Rating of Executive Functioning (D-REF)
Description: The Delis Rating of Executive Functioning (D-REF) contains 60 items rated by the parent to measure the child's executive functioning compared to age-peers. Results are calculated as T-scores, which have a mean of 50 and a standard deviation of 10. Here, we present the scores at study completion (visit 5), post-intervention. Greater values reflect greater executive functioning impairment.
Time Frame: D-REF will be administered at baseline and at the final visit (28 to 56 days after baseline). NOTE that baseline scores are listed previously in the appropriate section
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
t-score | 70.1 (11.9) | 73.2 (9.5)

8. Secondary Outcome: Change in Flanker Inhibitory Control and Attention Task
Description: The Flanker Inhibitory Control and Attention Task from the NIH Toolbox measure inhibitory control and attention. Task performance is in T-scores based on correct items and errors (mean of 50 and a standard deviation of 10). Here, we present difference scores between session 1 (baseline) T-score and 5 (completion) T-score. Greater values represents more change. Positive values represent improvement; negative values represent decline in performance.
Time Frame: NIH Toolbox will be administered at baseline and at the final visit (28 to 56 days after baseline)
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
Number analyzed (Participants) | 19 | 19
t-score | 2.05 (8.1) | 3.52 (8.92)

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Cognitive Training and Active tDCS | Cognitive Training and Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Training and Active tDCS (N=19) | Cognitive Training and Sham tDCS (N=19)
Headache (General disorders) | 5 (9) | 4 (4)
Scalp discomfort (Skin and subcutaneous tissue disorders) | 8 (19) | 7 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0)
Tingling (Skin and subcutaneous tissue disorders) | 6 (13) | 6 (6)
Itchiness (Skin and subcutaneous tissue disorders) | 8 (16) | 10 (13)
Sleepiness (General disorders) | 12 (31) | 12 (38)
Difficulty paying attention (General disorders) | 7 (10) | 5 (7)
Unusual feelings, attitudes, emotions (General disorders) | 2 (2) | 2 (2)
Tooth pain (General disorders) | 1 (2) | 0 (0)
Change in hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (8) | 0 (0)
Twitching / muscle movement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (3) | 0 (0)
Anxiety (General disorders) | 2 (7) | 1 (1)
Forgetfullness (General disorders) | 3 (3) | 3 (3)
Balance problem (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Change in dominant hand function (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT03361293/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03361293/ICF_001.pdf